CLINICAL TRIAL: NCT01304134
Title: A Prospective, Randomized, Blind, Multicentre, Parallel Group Study to Investigate the Efficacy and Safety of Oxycodone Hydrochloride Injection in the Postoperative Pain Relieving Treatment
Brief Title: Oxycodone Hydrochloride Injection in the Postoperative Pain Relieving Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OXYI09-CN-302
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Other Acute Postoperative Pain
MeSH Terms: interventions — Oxycodone; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxycodone i.v. (Experimental): To determine the efficacy and safety of oxycodone i.v. patient-controlled analgesia (PCA)
  Interventions: Drug: Oxycodone
- Morphine i.v. (Active Comparator): To determine the efficacy and safety of oxycodone i.v. patient-controlled analgesia (PCA)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Oxycodone — dosage:10mg/l dosage form:injection frequency:via PCA pump, background rate:0.5ml/h, 2ml/time duration:48 hours
  Other Names: Oxycodone Injection
  Arms: Oxycodone i.v.
Drug: Morphine — dosage: 10mg/ml dosage form: injection frequency: via PCA pump, background rate: 0.5ml/h, 2ml/times duration: 48 hours
  Other Names: Morphine Injection
  Arms: Morphine i.v.

SUMMARY:
To determine the efficacy and safety of oxycodone i.v. patient-controlled analgesia (PCA) in the pain relieving treatment during 48h postoperative period, by comparing with morphine i.v. PCA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged 18 to 65 years old, with a standard body weight [standard body weight = height (cm) - 100] ±15%.
2. ASA I and II.
3. Scheduled on elective open upper abdominal surgery under general anesthesia (liver, gall bladder, spleen, stomach, kidney, colon surgery), of which predicted operation duration is between 2-4h.
4. Hospitalized patients on non-emergency condition who have been given appropriate preoperative treatments.
5. Patients who are willing to participate in the study and have signed the written informed consent.
6. Negative pregnancy test result should be obtained for women of child-bearing age.

Exclusion Criteria:

1. Long-term analgesics or psychotropic drugs (including opioids, NSAIDs, sedatives, antidepressants) taken for the chronic pain, or patients abusing alcohol.
2. Body weight is less than or over ±15% of the standard body weight.
3. Severe impairment of liver and renal function at preoperative stage (ALT, AST, BUN, Cr).
4. Medical history of recovering from abnormal surgery anesthesia.
5. Medical history of hypertension (Systolic blood pressure ≥180Hg, Diastolic blood pressure 110Hg).
6. Esophagus reflux disease.
7. Sedatives, anti-emetics, and anti-pruritic drugs were taken 24 hours before operation.
8. Have known hypersensitivity to opioids.
9. Monoamine oxidase inhibitors and antidepressant drugs were taken within 15 days.
10. Patients with shock.
11. Patients with COPD.
12. Patients can not understand the VAS or unable to use PCA.
13. Pregnant or parturient women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Measuring VAS | 3h post-operation
  Measuring resting and coughing VAS, assessing the intensity of pain
Measuring VAS | 24 hours post operation
  Measuring resting and coughing VAS, assessing the intensity of pain
Measuring VAS | 48 hours post operation
  Measuring resting and coughing VAS, assessing the intensity of pain

SECONDARY OUTCOMES:
Dosage | Within 48h
  Total dosage of study drugs within 48h.
The dosage of other rescue analgesic drugs used within 48h post-operation. | 48hrs
  The dosage of other rescue analgesic drugs used within 48h post-operation.
The invalid times and the total times of PCA application | 48hrs
  The invalid times and the total times of PCA application
Satisfaction degree for analgesia | 48hrs
  Satisfaction degree for analgesia after the treatment
AE occurrence and abnormal lab value | 48hrs
  AE and normal lab value will be recorded during the study

CONTACTS AND LOCATIONS:
Overall Officials: Mundipharma China Ltd., Study Chair — Mundipharma China Ltd.; Mundipharma China Ltd., Principal Investigator — Investigational Site Beijing, China
Locations (1):
- Investigational site, Beijing, Beijing Municipality, China